CLINICAL TRIAL: NCT04514744
Title: Dynamic Proteomics and Integrated Rates of Muscle Protein Synthesis During an Acute Period of Hypertrophy and Atrophy (HYPAT) in Young, Healthy Men
Brief Title: Dynamic Proteomics and Integrated Rates of Muscle Protein Synthesis During an Acute Period of Loading and Unloading
Acronym: HYPAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10624
Record Dates: First submitted 2020-06-29; First posted 2020-08-17 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Proteomics; Exercise; Atrophy, Disuse; Hypertrophy
MeSH Terms: conditions — Motor Activity; Muscular Disorders, Atrophic; Hypertrophy

STUDY DESIGN:
Intervention Model Description: In a randomized fashion, one participant will have one leg assigned to unilateral immobilization, and the other leg will undergo unilateral resistance exercise training, for 8 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Immobilization (Experimental): One leg will undergo 14 days of single-leg immobilization, by means of a removable knee brace.
  Interventions: Procedure: Knee bracing
- Unilateral Resistance Exercise (Experimental): One leg will undergo 4 sessions of unilateral resistance exercise, over the course of 8 days. Specifically, participants will be asked to perform leg press and leg extension.
  Interventions: Other: Unilateral Resistance Exercise Training

INTERVENTIONS:
Procedure: Knee bracing — Participants will have one leg immobilized, by means of a removable Don Joy Knee Brace. Participants will be expected to keep the knee brace on for 14 days, completely prevent weight bearing on the immobilized leg, and use crutches.
  Arms: Unilateral Immobilization
Other: Unilateral Resistance Exercise Training — Participants will perform resistance training on 4 occasions throughout an 8 day time period.
  Arms: Unilateral Resistance Exercise

SUMMARY:
Skeletal muscle plays several different roles in the promotion and maintenance of health and well-being. The loss of muscle mass that occurs with aging, chronic muscle wasting diseases, and physical inactivity puts people at an increased risk of frailty and becoming insulin resistant, and therefore imposes a significant burden on health care spending. Resistance exercise participation has proven particularly effective for increasing muscle mass and strength. This effectiveness can be used by health care practitioners in a rehabilitation setting to promote the recovery of individuals who have undergone involuntary periods of muscular unloading (i.e. limb immobilization caused by a sports injury or reconstructive surgery). However, there is large variability in the amount of muscle mass and strength that people gain following participation in resistance exercise. Some individuals fail to increase the size of their muscle (low responders) whereas others show vary large increases in muscle size (high responders) in response to the same resistance training program. People also show differences in the amount of muscle tissue they lose when they have a limb immobilized. To circumvent variability across individuals, the investigators utilized a within-person paired Hypertrophy and Atrophy ('HYPAT') strategy that reduced response heterogeneity by ~40% (Available at: https://ssrn.com/abstract=3445673). Specifically, one leg performed resistance training for 10 weeks to induce hypertrophy, whereas the other leg underwent single-leg immobilization for 2 weeks to induce atrophy. The primary goal of the study will be to gain insight into the molecular responses to an acute period of single-leg immobilization and resistance exercise (8 days). The investigators will use an integrated systems biology approach to monitor the individual rates of over one hundred different muscle proteins.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, between the ages of 18 and 30 y
* Body Mass Index between 18.5 and 30.0 kg/m2
* Able and willing to provide informed consent

Exclusion Criteria:

* A history of neuromuscular disorders or muscle/bone wasting diseases.
* Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin-dependent or insulin-independent diabetes, or the presence of any other metabolic disease - all of which will be determined via a medical history screening questionnaire.
* The use of any medications known to affect protein metabolism (glucocorticoids, non-steroidal anti-inflammatory medication, or prescription strength acne medication, etc.).
* A (family) history of thrombosis.
* The use of anticoagulant medications.
* Consumption of tobacco-containing products.
* Excessive alcohol consumption (>21 units/wk).
* History of bleeding diathesis, platelet or coagulation disorders, or anti-platelet/anticoagulation therapy.
* Exercise participation >2 days/wk (structured resistance and/or aerobic-type exercise)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dynamic Proteomics | Baseline, Day 5, Day 9 and Day 14 (Post)
  The investigators will use deuterated water and skeletal muscle biopsies, paired with sensitive Gas Chromatography-Mass Spectrometry techniques to calculate the individual synthesis rate of over one hundred different skeletal muscle proteins.
Change in Integrated Rates of Muscle Protein Synthesis | Baseline, Day 5, Day 9 and Day 14 (Post)
  The investigators will use deuterated water and skeletal muscle biopsies to calculate the cumulative synthesis of skeletal muscle proteins.

SECONDARY OUTCOMES:
Change in Lean Mass Using Dual X-Ray Absorptiometry | Baseline, Day 5 and Day 14 (Post)
  The change in lean mass (kg) will be assessed throughout the intervention using dual X-Ray absorptiometry at baseline, Day 4, and Day 8 (Post) of the intervention
Change in Muscle Strength using an Isokinetic Dynamometer | Baseline, Day 5 and Day 14 (Post)
  Muscle strength will be analyzed throughout the intervention using an isokinetic dynamometer. Isometric muscle torque (i.e., strength [N*m]) of the knee extensor will be measured.
Change in Muscle Cross-Sectional Area using Ultrasonography | Baseline, Day 5 and Day 14 (Post)
  The investigators will measure changes in vastus lateralis muscle cross sectional area (cm^2) throughout the intervention using ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All participants will be assigned a unique subject ID, and therefore, other researchers involved with analyses will not have access to identifying participant information.